CLINICAL TRIAL: NCT03227744
Title: A Pilot Study of Prostate Cancer-specific Anxiety in Active Surveillance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been terminated
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17314
Record Dates: First submitted 2017-06-30; First posted 2017-07-24 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer, Anxiety
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders | interventions — Psychotherapy, Group; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enrolled in group therapy (Active Comparator): Patients in the group therapy arm will be enrolled in group therapy and be issued surveys.
  Interventions: Behavioral: Group therapy; Other: Surveys
- Not enrolled in group therapy (Placebo Comparator): Patients in control arm will be issued surveys
  Interventions: Other: Surveys

INTERVENTIONS:
Behavioral: Group therapy — Twelve 1-hour group therapy sessions with a licensed psychologist for prostate-cancer related anxiety.
  Arms: Enrolled in group therapy
Other: Surveys — MAX-PC, GAD and FACT-P

SUMMARY:
This study is a clinical trial to determine whether a 12-week group therapy intervention for patients undergoing Active Surveillance for Prostate Cancer can relieve disease-related anxiety and improve quality of life and delay elective treatment of prostate cancer. The goal of the study is to further our understanding of anxiety in men who have been diagnosed with prostate cancer and are undergoing Active Surveillance. Men who have elected Active Surveillance for their management of prostate cancer are eligible to participate in this study. After signing informed consent, all participants will complete two brief questionnaires (The Memorial Anxiety Scale for Prostate Cancer [MAX-PC] and the General Anxiety and Depression Scale 7 [GAD-7] to measure their anxiety levels. If the participant scores above a certain number, they will be asked to participate in the study. Patients will be randomly assigned to either a control group, who will receive no treatment, but continue to follow up with their urologist to manage their prostate cancer as usual, or the treatment group. The treatment group will receive 12 one-hour group therapy sessions that will take place once a week for 12 weeks with a licensed psychologist free of charge. They will be instructed to follow up with their urologist as previously determined for their prostate cancer management. Patients in both groups will be monitored for anxiety completing three questionnaires, the MAX-PC and GAD-7 which they previously completed, and the Functional Assessment of Cancer Therapy - Prostate (FACT-P) during the 4th and 12th weeks of therapy. If patients require further therapy beyond the group treatment sessions, the investigators may refer them to a psychologist or psychiatrist for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40
* Primary diagnosis of Prostate Cancer
* Initial MAX-PC score of ≥16.
* Sign a consent form allowing related information to be included in this research.

Exclusion Criteria:

* Prostate cancer is not their primary diagnosis.
* Have pre-existing diagnosed psychiatric conditions, are currently taking psychotropic medications (e.g., antidepressants, anxiolytics, mood stabilizers.)
* Have been diagnosed with cancer other than prostate cancer (and non-melanoma skin cancer)
* Evidence of active substance abuse.
* Participants in the treatment group who are absent from more than 3 therapy sessions will be excluded.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Assessment of MAX-PC Scores | Change from baseline to 4 weeks to 12 weeks
  Two groups, the experimental (recipients of group therapy) and the control (literature only) will be compared for anxiety based on their MAX-PC questionnaire scores. Eighteen questions about anxiety related to prostate cancer and prostate specific antigen (PSA) tests are graded from 0-3 (0 = not at all; 3 = often), yielding a total between 0 and 54.
Assessment of FACT-P Scores | Change from baseline to 4 weeks to 12 weeks
  Two groups, the experimental (recipients of group therapy) and the control (literature only) will be compared for anxiety based on their FACT-P questionnaire scores. Twenty-seven questions about physical, social/family, emotional and functional well-being are graded from 0-4 (0 = not at all; 4 = very much), yielding a total between 0 and 108.

SECONDARY OUTCOMES:
Assessment of anxiety scores as a function of time | Change from baseline to 4 weeks to 12 weeks
  In secondary analysis, a mixed effects model will be used when the outcome vector consists of all three measurements (baseline, 4 and 12 weeks) and via statistical contrasts will examine whether the relationship between PSA anxiety scores and time is linear or if the effect of intervention on anxiety scores is fully observed by week 4. Two-sided p-values ≤ 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Pinkhasov, MD, Principal Investigator — NYU Winthrop Hospital
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

DOCUMENTS (2):
  • Study Protocol (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03227744/Prot_000.pdf
  • Informed Consent Form (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03227744/ICF_001.pdf